CLINICAL TRIAL: NCT05026593
Title: A Randomized, Multicenter, Open-Label, Phase Ib Study to Evaluate Efficacy, Safety and Tolerability of IBI110 in Combination With Sintilimab Plus Etoposide and Platinum or Carboplatin in Patients With Untreated Extensive-Stage Small Cell Lung Cancer
Brief Title: A Study of IBI110 in Combination With Sintilimab and Chemotherapy in Patients With Untreated Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI110A201
Record Dates: First submitted 2021-08-16; First posted 2021-08-30 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2022-07

CONDITIONS: SCLC
MeSH Terms: interventions — Carboplatin; Cisplatin; Etoposide; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sintilimab+EP (Active Comparator): During each 21-day cycle, participants receive Sintilimab 200 mg intravenously (IV) Day 1 PLUS etoposide 100 mg/m^2 IV on Days 1, 2 and 3 PLUS investigator's choice of platinum (carboplatin titrated to an area under the plasma drug concentration-time curve [AUC] 5 IV on Day 1 OR cisplatin 75 mg/m^2 IV on Day 1). After the induction phase, participants will begin maintenance therapy with Sintilimab 200 mg intravenously (IV) Day 1 every 3 weeks until PD, unacceptable toxicity, withdrawal of consent, or other protocol-allowed reasons, whichever occurs first.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide; Drug: Sintilimab
- IBI110+Sintilimab+EP (Experimental): During each 21-day cycle, participants receive IBI110 PR2D intravenously (IV) Day 1 PLUS Sintilimab 200 mg intravenously (IV) Day 1 PLUS etoposide 100 mg/m^2 IV on Days 1, 2 and 3 PLUS investigator's choice of platinum (carboplatin titrated to an area under the plasma drug concentration-time curve [AUC] 5 IV on Day 1 OR cisplatin 75 mg/m^2 IV on Day 1). After the induction phase, participants will begin maintenance therapy with IBI110 PR2D intravenously (IV) Day 1 PLUS Sintilimab 200 mg intravenously (IV) Day 1 every 3 weeks until PD, unacceptable toxicity, withdrawal of consent, or other protocol-allowed reasons, whichever occurs first.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide; Drug: Sintilimab; Drug: IBI110

INTERVENTIONS:
Drug: Carboplatin — Carboplatin will be administered after completion of Sintilimab by IV infusion to achieve an initial target AUC of 5 mg/mL/min on Day 1.
Drug: Cisplatin — Cisplatin 75 mg/m^2 will be administered after completion of Sintilimab by IV infusion on Day 1.
Drug: Etoposide — Etoposide 100 mg/m^2 will be administered by IV infusion following carboplatin or cisplatin administration, during the induction phase on Day 1 through 3 of each cycle. On Days 2 and 3, patients will receive etoposide alone.
Drug: Sintilimab — Sintilimab 200 mg will be administered by IV infusion following IBI110 on Day 1 of each 21-day .
Drug: IBI110 — IBI110 RP2D will be administered by IV infusion on Day 1 of each 21-day .
  Arms: IBI110+Sintilimab+EP

SUMMARY:
IBI110 is an investigational drug under evaluation for treatment of small cell lung cancer. The purpose of the study was to assess the Efficacy and Safety of IBI110 in combination with Sintilimab and chemotherapy with untreated ES-SCLC.

DETAILED DESCRIPTION:
This Phase II, multicenter, open-lable study is designed to evaluate the safety and efficacy of IBI110 (anti-lymphocyte activation gene 3 [LAG-3] monoclonal antibody) and sintilimab (anti-programmed death 1 [PD-1] antibody) in combination with intravenous (IV) cisplatin/carboplatin plus (+) etoposide (EP) in treatment naïve patients with extensive-stage small cell lung cancer (ES-SCLC) . Sixty eligible subjects will be enrolled and randomized in a 1:1 ratio to the experimental arm or the control arm. The experimental arm will be IBI110+ sintilimab + EP Q3W for 4 cycles, followed by IBI110+ sintilimab Q3W until disease progression. The control arm will be sintilimab + EP Q3W for 4 cycles, followed by sintilimab Q3W until disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have the ability to understand and voluntarily sign informed consent;
2. Age: over 18 years old;
3. Expected survival period ≥ 3 months;
4. Histologically or cytologically confirmed ES-SCLC (according to the Veterans Lung Administration Lung Study Group, VALG staging);
5. No prior systemic treatment for ES-SCLC;
6. Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1;
7. At least 1 measurable lesion by computed tomography (CT) or magnetic resonance imaging (MRI) per Response Eval -uation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria;
8. Adequate hematologic and end organ function.

Exclusion Criteria:

1. Have been previously exposed to any antibody or drug of immune-mediated therapy, including but not limited to LAG-3, anti-cytotoxic T lymphocyte antigen-4 (CTLA-4), anti-PD-1, anti-PD-L1 antibodies.
2. Have received systemic treatment with Chinese herbal medicine or immunomodulatory drugs with anti-tumor indications (including thymosin, interferon, interleukin, except for local use to control pleural effusion) within 2 weeks prior to the first administration of study drug.
3. Have active or uncontrolled central nervous system (CNS) metastases and/or spinal cord compression and/or carcinomatous meningitis, or history of leptomeningeal carcinoma. Subjects with a history of radiotherapy or surgery for brain metastases and asymptomatic CNS metastases at the time of screeing are eligible if they meet all of the following criterias: have measurable lesions outside the CNS; do not have midbrain, pons, meninges, medulla oblongata or spinal cord metastases; do not have evidence of new or enlarged brain metastases after treatment for brain metastases, and corticosteroids and anticonvulsants treatments have been discontinued for at least 14 days prior to the study treatment. Subjects with asymptomatic brain metastases can be included if the brain metastases have been treated with radiotherapy and above mentioned criterias are all met.
4. Are expected to require any other antineoplastic therapy while in study (PCI is allowed).
5. Have received administration of live attenuated vaccines within 4 weeks prior to the first administration of study drug or anticipation that such a live attenuated vaccine will be required during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 5 years
  PFS is defined as the time interval from ra ndomization to the date of the first docu mented tumor progression, based on inve stigator assessments (per RECIST 1.1), or death due to any cause, whichever come s first.
Incidence of Treatment-related Adverse Events(TRAE), Serious Adverse Events (SAEs) and Immune-related adverse events (irAE) nation with sintilimab and EP in untreated ES-SCLC | Up to 5 years
  Evaluate the safety and tolerability profile of IBI110 + sintilimab and EP in untreated ES-SCLC . Adverse events per CTCAE v5.0 criteria guidelines will be used to assess this outcome.

SECONDARY OUTCOMES:
Overall Survival(OS) | Up to 5 years
  OS: Defined as the time interval from ran domization to death.
Objective response rate(ORR) | Up to 5 years
  ORR: Defined as the number of cases achi eving CR, or PR, as a percentage of patien ts with evaluable efficacy.
Disease control rate(DCR); | Up to 5 years
  DCR: The percentage of cases that achiev ed remission (PR+CR) and stable disease (SD) after treatment accounted for the n umber of evaluable cases.
Duration of response(DOR); | Up to 5 years
  DOR: Defined as the time from the first d ocumented objective response to the first documented progressive disease or deat h of any cause, whichever occurs first.
To assess the immunogenicity; | Up to 5 years
  Immunogenicity: the immunogenicity: will be evaluated by determining the inciden ce of anti-drug antibodies (ADA) and furt her testing ADA-positive serum specimen s for neutralizing antibody (Nab);
To assess the Area under the plasma concentration versus time curve(AUC) of IBI110+Sintilimab+EP | Up to 1 year
To assess the Peak Plasma Concentration(Cmax) of IBI110+Sintilimab+EP | Up to 1 year
To assess the half-life(t1/2) of IBI110+Sintilimab+EP | Up to 1 year
To assess the clearance(CL) of IBI110+Sintilimab+EP | Up to 1 year
To assess the volume of distribution(V) of IBI110+Sintilimab+EP | Up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China